CLINICAL TRIAL: NCT05239624
Title: Enfortumab Vedotin in Combination With Pembrolizumab for Locally Advanced and/or Node Positive Urothelial Carcinoma Prior to Surgery (EV-ECLIPSE)
Brief Title: Enfortumab Vedotin and Pembrolizumab in People With Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); Seagen Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-316
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
Keywords: Locally Advanced and/or Node Positive; Enfortumab vedotin; Pembrolizumab; Clinical Stage T2-T4, N1-N3, M0 OR cT1, N2-N3, M0; 21-316
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a phase II trial of enfortumab vedotin in combination with pembrolizumab as first-line therapy for patients with locally-advanced or node positive urothelial carcinoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- enfortumab vedotin in combination with pembrolizumab (Experimental): Enfortumab vedotin will be administered at 1.25 mg/kg on day 1 and day 8 of each 21-day cycle, for up to 6 cycles. Patients can proceed to surgery prior to completion of cycle 6 at the discretion of the investigator and urologist if toxicities prevent completion of 6 cycles of treatment. Enfortumab vedotin will be capped at a maximum dose of 125 mg for each infusion (for patients who weigh > 100 kg). Pembrolizumab will be administered on day 1 of each cycle, every 21 days, for 6 cycles. After completion of 3 cycles patients with have imaging assessment, and patients with progression of disease as measured by distant metastases will be removed from the study. At completion of cycle 6, patients will have repeat imaging assessment and proceed to cystectomy within 4-8 weeks. Following cystectomy, patients will resume pembrolizumab monotherapy on day 1 of each 21-day cycle for an additional 11 doses (Cycles 7-17), to complete 1 year of pembrolizumab therapy.
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — Enfortumab vedotin will be administered at 1.25 mg/kg on day 1 and day 8 of each 21-day cycle, for up to 6 cycles.
Drug: Pembrolizumab — Pembrolizumab will be administered on day 1 of each cycle, every 21 days, for 6 cycles.

SUMMARY:
This study will test whether enfortumab vedotin combined with pembrolizumab is an effective treatment for people with bladder cancer (urothelial carcinoma) involving the lymph nodes who are going to have surgery to remove their cancer (cystectomy). The researchers will look at whether treatment with enfortumab vedotin and pembrolizumab before surgery can get rid of cancer within the lymph nodes. They will also try to find out if this combination of drugs is effective at shrinking participants' cancer before their surgery.

The researchers think that a combination of enfortumab vedotin and pembrolizumab may help people with this disease because both drugs are designed to help the immune system attack and kill cancer cells. The researchers think the drugs may be more effective if given in combination rather than on their own.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of muscle invasive bladder cancer (previously known as transitional cell) carcinoma (i.e., cancer of the bladder, renal pelvis, ureter, or urethra)
* Clinical Stage T2-T4, N1-N3, M0 OR cT1, N2-N3, M0
* Pathology:

  * Representative urothelial carcinoma FFPE tumor specimens (tumor blocks or 20 unstained slides). Patients with < 20 slides may be enrolled after discussion with the principal investigator.
  * Muscle invasive urothelial carcinoma of the bladder histologically confirmed at the enrolling institution from TURBT. (Urothelial carcinoma invading into the prostatic stroma with no histologic muscle invasion is allowed provided the extent of disease is confirmed via imaging and/or EUA.)
  * Evidence of urothelial carcinoma from FNA of lymph node OR lymphadenopathy suspicious for nodal disease on cross-sectional imaging, MRI, or u/s.
  * Node positivity for eligibility will be defined as imaging read with suspicious lymph node ≤ 1.0 cm in the short axis, with biopsy, as documented by the radiologist at the treating center. While biopsy to confirm lymph node involvement is preferred, patients without biopsy proven urothelial carcinoma in lymph nodes may be enrolled if imaging shows a lymph node ≥ 1.0 cm in the short axis, and with confirmation from the study principal investigator. If biopsy positive, LN can be any size. If biopsy not performed, LN ≥ 1.0 cm in short axis.
* Deemed medically appropriate for radical cystectomy with treatment response achieved, as per MSK or participating site Attending Urologic Oncologist
* Platinum eligible and ineligible patients are permitted on study
* No prior treatments for muscle invasive or metastatic urothelial carcinoma
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Estimated glomerular filtration rate (eGFR) ≥ 30 ml/min/1.73 m2 using the CKD-EPI equation: eGFR = 141 x min(Scr/k, 1)a x max (Scr/k, 1)-1.209 x 0.993Age x 1.018 [if female] x 1.159 [if black]

  °Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1
* Be willing and able to provide written informed consent for the trial
* Contraception requirements:

  1. Male participants:

     A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days following the last dose of treatment, corresponding to time needed to eliminate any study treatment(s) (e.g. 5 terminal half-lives for pembrolizumab and enfortumab vedotin) plus an additional 90 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period.
  2. Female participants:

A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

i. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR ii. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least [90 days (corresponding to time needed to eliminate any study treatment(s) (pembrolizumab and enfortumab vedotin) plus 30 days (a menstruation cycle)] after the last dose of study treatment.

* Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 14 days prior to the start of study treatment either prior to consent or at the study screening visit.
* Hematological

  * Absolute neutrophil count (ANC) ≥1500/μL
  * Platelets ≥100 000/μL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
* Renal

  °Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) GFR or CrCl of ≥ 30 mL/min
* Hepatic

  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN
* Coagulation °International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks. b eGFR as calculated by the CKD-EPI equation can be used in place of the creatinine clearance

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies

Exclusion Criteria:

* Evidence of NYHA functional class III or IV heart disease
* Any of the following within 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* On-going cardiac dysrhythmias of NCI CTCAE Version 5.0 grade ≥ 2. However, stable atrial fibrillation controlled medically or with a device (i.e. pacemaker) or prior ablation is allowed
* Pre-existing sensory grade ≥ 2 neuropathy
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure aside from cystectomy during the course of the study. Transurethral resection or other urinary tract diagnostic procedures, excisional biopsy, IR-guided biopsy, or MEDIPORT placement are NOT defined as major surgical procedures.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

* Is currently enrolled in another therapeutic trial. Patients cannot receive concurrent treatment on another clinical trial; Patients are allowed to enroll on supportive care trials or non-treatment trials (e.g. QOL, dietary survey studies) concurrently
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

  * Prior treatment with an antibody drug conjugate for bladder cancer directed therapy
  * Prior systemic chemotherapy (prior intravesical therapy is allowed)
  * Prior radiation therapy to the bladder
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. 1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Administration of killed vaccines is allowed. COVID-19 vaccination is permitted.

  °Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Has receieved intravesical bacillus Calmette-Guerin (BCG) within 4 weeks before Cycle 1, Day 1 14.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a history of poorly controlled human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) related illness. Patients with a history of an aids-defining opportunistic infection within the last 12 months or who are on prophylactic antimicrobials related to underlying HIV are not eligible. Patients with a history of HIV and a CD4 T cell count of ≥350 are eligible to enroll in this study with the approval of the study PI.
* Subjects with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Has a history of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, vascular thrombosis associated with antiphospholipid syndrome, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, systemic vasculitis, or glomerulonephritis.

  * Patients with history of autoimmune related hypothyroidism on stable dose of thyroid replacement hormone may be eligible for this study
  * Patients with controlled Type I diabetes mellitus on a stable dose of insulin may be eligible for this study
* Has a history of idiopathic pulmonary fibrosis, pneumonitis/interstitial lung disease that requires steroids or has current pneumonitis/interstitial lung disease (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Patients with active hepatitis B virus (HBV, chronic or acute, defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C antibody

  * Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to Cycle 1, Day 1 and confirmed to be negative.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active tuberculosis or BCG infection
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1. Abnormal urinalysis does not constitute signs/symptoms of infection unless urine culture obtained at screening grows ≥ 100,000 colonies of bacteria.
* Therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1

  * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
  * Patients receiving antibiotics for active infection are not eligible
* Prior allogeneic stem cell or solid organ transplant
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia
* Patients with a history of or active bone marrow disorders expected to interfere with study therapy (e.g. acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma)
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; and inherited liver disease
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Patients with active keratitis or history of corneal ulcers are excluded
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-ofcare management (e.g. prostate cancer with Gleason score ≤ 7, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR Rate) | 2 years
  Defined as lack of muscle invasive carcinoma (<pT2) and the absence of lymph node metastasis (N0) in the final cystectomy specimen. Pathologic complete response to perioperative treatment is defined as the absence of carcinoma (pT0) and the absence of lymph node metastases (N0). Pathologists will assess surgical specimens systematically using criteria agreed upon for all conventional neoadjuvant treatment based on the AJCC TNM staging system.

SECONDARY OUTCOMES:
Event free survival (EFS) | 2 years
  Event-free survival will be measured from the initiation of treatment. Any of the following events will qualify as an event:
  * Primary progression of disease (from time of confirmatory scan)
  * Recurrence of disease post-operatively with metastatic or local pelvic recurrence after radical cystectomy.
  * Patients who do not proceed to cystectomy due to toxicity
  * The assessment of disease recurrence versus development of a second primary tumor will be left to the discretion of the treating physician. If the patient did not progress nor die, the patient will be censored on the date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Aggen, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering -Nassau, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York
  - Lehigh Valley Health Network (Data Collection Only), Allentown, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm